CLINICAL TRIAL: NCT00766870
Title: A Randomised, Double-blind, Parallel-group, Placebo-controlled, and Active-referenced Study Evaluating the Efficacy and Safety of Three Fixed Dose Regimens of Lu AA34893 in the Treatment of Major Depressive Disorder
Brief Title: Efficacy and Safety of Lu AA34893 in Patients With Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was previously paused and is now terminated
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12279A; 2007-007025-51 (EudraCT Number)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Major Depressive Disorder
Keywords: Efficacy; Safety; Depression; Interventional; Placebo; Short-term; Major Depressive Disorder; Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Lu AA34893
- 2 (Experimental)
  Interventions: Drug: Lu AA34893
- 3 (Experimental)
  Interventions: Drug: Lu AA34893
- 4 (Other)
  Interventions: Drug: Venlafaxine extended release
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA34893 — Per oral doses, divided in twice daily administrations as capsules during 8 weeks, followed by a two-week tapering period
  Arms: 1; 2; 3
Drug: Venlafaxine extended release — Per oral, once daily, during 8 weeks, followed by a two-week tapering period
  Arms: 4
Drug: Placebo — Per oral doses, twice daily as capsules during 10 weeks
  Arms: 5

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety and tolerability of three fixed dosages of Lu AA34893 compared to placebo in the treatment of patients with Major Depressive Disorder.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is reported to be the most common mood disorder, with a lifetime prevalence of about 15% and as high as 25% in women. MDD is characterised by the presence of one or more Major Depressive Episodes (MDEs) that presents with depressed mood, loss of interest or pleasure, disturbed sleep or appetite, low energy, feelings of guilt or low self-worth, and poor concentration. MDD is a disabling, severe illness that tends to be chronic, and repeated episodes are common. Despite the availability of a range of effective treatments in MDD, a significant proportion of patients do not respond or achieve remission and many relapse despite continued treatment. Lu AA34893 has a novel mechanism of action and this could be of clinical relevance in addressing currently unmet needs in MDD.

ELIGIBILITY:
In- and out-patients with moderate to severe Major Depressive Disorder

Inclusion Criteria:

* Major Depressive Episode (MDE) as primary diagnosis according to DSM-IV (classification code 296.xx)
* Moderate to severe depression
* Current MDE duration of at least 3 months

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the DSM-IV TR
* Any substance disorder within the previous 6 months
* Females of childbearing potential and not using adequate contraception
* Use of any psychoactive medication within 2 weeks before randomisation and during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured by the change from baseline in MADRS total score | 8 weeks

SECONDARY OUTCOMES:
HAM-D, CGI, responders and remitters, HAM-A, adverse events, clinical safety laboratory tests, vital signs, weight, ECG, physical examination | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CA009, Mississauga, Ontario, Canada